CLINICAL TRIAL: NCT06592859
Title: Quzhou Population Cohort Research Project (Aging Related Research: Intervention of Nicotinamide Mononucleotide in Middle-aged and Elderly People)
Acronym: NMNAGING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: People's Hospital of Quzhou (Other)
Collaborators: Beijing Institute of Genomics, Chinese Academy of Sciences (Other Government); Institute of Zoology, Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Feng Zhang, researcher, People's Hospital of Quzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-049; MR-33-24-001563 (Other: Medical Research Registration and Filing Information System)
Record Dates: First submitted 2024-07-30; First posted 2024-09-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-09

CONDITIONS: Aging; NMN
Keywords: Aging; NMN

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMN Arm (Experimental): NMN Arm participants took one capsule (containing 350mg NMN) with breakfast daily for one year.
  Interventions: Dietary Supplement: NMN
- Placebo Arm (Placebo Comparator): Placebo arm participants took one capsule (appearance and odor are the same as NMN) with breakfast daily for one year.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: NMN — NMN Arm participants took one capsule (containing 350mg NMN or placebo) with breakfast daily for one year.
  Arms: NMN Arm
Dietary Supplement: placebo — Placebo arm participants took one capsule (appearance and odor are the same as NMN) with breakfast daily for one year.
  Arms: Placebo Arm

SUMMARY:
This study is a single center, randomized, double-blind, placebo-controlled clinical trial of drug intervention on aging. The purpose is to explore the effectiveness of NMN on the premise of ensuring the safety of oral drug, in order to provide effective intervention means for delaying aging and improve the quality of life of the elderly population. The main outcome measures of this study were the efficacy and safety of NMN on aging intervention.

ELIGIBILITY:
Inclusion criteria：

1. Local residents of Quzhou or living in Quzhou for over ten years.
2. age 40-50 and 60-70 years old, no major bad habits.
3. Gender unlimited.
4. in good health and has not undergone major surgery within half a year.
5. Be able to communicate well with researchers and cooperate with the work during the study.
6. Written informed consent can be signed voluntarily.

Exclusion criteria：

1. Alcoholism, heavy smoking (more than 5 packs/day, 20 cigarettes per pack), drug abuse or substance abuse.
2. Participants are conducting other clinical trials or using any research drugs or equipment for treatment within 30 days before enrollment (including but not limited to aspirin, metformin, resveratrol, vitamin C, etc.).
3. Obesity (bmi more than 30).
4. Pregnant/lactating women.
5. Disease history:

   A) under 60 years old:
   1. any cancer (erythrocytosis, except basal cell or squamous cell skin cancer).
   2. coronary artery disease/myocardial infarction/clinically significant congestive heart failure.
   3. stroke/transient ischemic attack.
   4. deep vein thrombosis/pulmonary embolism.
   5. serum creatinine > 1.5 mg/dl (male).
   6. poor control of hypertension (although treated, there is still significant hypertension (systolic blood pressure > 160 mmHg, or diastolic blood pressure >100 mmHg)).
   7. history of active liver disease or metabolic acidosis.
   8. chronic kidney disease/hemodialysis treatment, history of severe kidney damage and/or EGFR ≤ 45ml/min/1.73m2.
   9. severe autoimmunity/inflammation, such as rheumatoid arthritis, lupus, Crohn's disease, etc.
   10. nervous system diseases such as dementia, such as Alzheimer/Parkinson's disease.
   11. diabetes mellitus (hemoglobin > 6.5% or fasting blood glucose > 126 mg/dL or taking diabetes drugs or insulin treatment).
   12. recent (within 3 months) cardiovascular events (myocardial infarction, coronary intervention, coronary artery bypass grafting).
   13. infectious diseases such as HIV, hepatitis, tuberculosis, etc.
   14. hand or lower limb disability affects normal function and life.

   B) older than 60 years:
   1. any cancer (erythrocytosis, except basal cell or squamous cell skin cancer).
   2. history of active liver disease or metabolic acidosis.
   3. chronic kidney disease/hemodialysis treatment, history of severe kidney damage and/or EGFR ≤ 45ml/min/1.73m2.
   4. severe autoimmunity/inflammation, such as lupus, Crohn's disease, etc.
   5. nervous system diseases such as dementia, such as Alzheimer/Parkinson's disease.
   6. recent (within 3 months) cardiovascular events (myocardial infarction, coronary intervention, coronary artery bypass grafting).
   7. infectious diseases such as HIV, hepatitis, tuberculosis, etc.
   8. hand or lower limb disability affects normal function and life.
6. Currently taking the following drugs regularly:

   A) chemotherapy drugs (such as tamoxifen, adriamycin, mitoxantrone, bleomycin). B) antiplatelet drugs (e.g., clopidogrel/Plavix, dipyridamole/anglionide, ticlopidine/ticlopidine, except aspirin).

   C) cholinesterase inhibitors for Alzheimer's disease (donepezil/alicept).
7. The researchers believe that the physical factors of the participants may have an adverse impact on the research process or results.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
blood NAD+ levels | Baseline, 6 months and 12 months
  NAD+ concentration in serum
SF-36 questionnaire | Baseline, 6 months and 12 months
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.

SECONDARY OUTCOMES:
bone density | Baseline, 6 months and 12 months
  Bone density of the lumbar spine will be measured by using dual-energy X-ray absorptiometry.
FVC | Baseline, 6 months and 12 months
  forced vital capacity will be measured by pulmonary function test.
FEV1 | Baseline, 6 months and 12 months
  Forced expiratory volume in one second will be measured by pulmonary function test.
grip strength test | Baseline, 6 months and 12 months
  One handed grip strength test is used to evaluate physical strength.
flexibility of fingers | Baseline, 6 months and 12 months
  Purdue Pegboard Test is used to test the flexibility and coordination of participants. Participant is required to insert as many pegs as possible into the board in one minute. The number of insertions is considered an indicator of flexibility.

OTHER OUTCOMES:
BMI | Baseline, 6 months and 12 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
blood pressure | Baseline, 6 months and 12 months
  Measuring blood pressure at rest.
Changes in the body composition | Baseline, 6 months and 12 months
  Fat mass, muscle mass, visceral fat, water mass determined by Bioelectrical Impedance Analysis (BIA).

CONTACTS AND LOCATIONS:
Locations (1):
- People's Hospital of Quzhou, Quzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No